CLINICAL TRIAL: NCT05171452
Title: Proof-of-concept Study to Assess Urinary PGE-MUM Concentration (PROSTAGLANDIN E-MAJOR URINARY METABOLITE) as a Potential Marker of Inflammation in Inflammatory Bowel Disease (IBD) - Comparison With Fecal Calprotectin Level (FC)
Brief Title: Urinary PGE-MUM (PROSTAGLANDIN E-MAJOR URINARY METABOLITE) as Inflammatory Marker in Chronic Inflammatory Bowel Disease
Acronym: MICIMUM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180450; 2018-A02342-53 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2021-12-10; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory bowel diseases; urinary marker
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Adult IBD with active inflammation
  Interventions: Biological: Urine and stoll samples
- Group B: Adult IBD in remission
  Interventions: Biological: Urine and stoll samples

INTERVENTIONS:
Biological: Urine and stoll samples — Urine collection will be proposed to patient during consultations or medical examinations corresponding to routine care of patients with IBD at the time of prescribing a FC test. The urine sample, as for stool samples, will be collected in an ordinary universal container at any time of the day (no dietary restriction is required). Urine and stool samples should be taken during the same period (for example, the same day, or within a maximum of one week if no change in treatment)

SUMMARY:
The inflammatory bowel diseases (IBD) are lifelong, relapsing-remitting diseases. As the timing of relapse is unpredictable, and current monitoring is symptoms-based, there remains a window between the initial upregulation of the inflammatory response and the onset of clinical symptoms at which point the inflammatory episode is well established. The use of endoscopy as means of predicting relapse is not suitable for regular use. The potential role of Fecal calprotectin (FC) in IBD in predicating the risk of relapse has been well investigated with key studies. Its fecal concentration is proportional to neutrophilic influx into the intestinal tract, which is a feature of active IBD. FC correlates well with the severity of endoscopic lesions. After excretion, FC remains stable in the feces for 1 week at room temperature. However, its considerable daily variation suggests interfering factors discrete from inflammatory disease. There is increasing research into novel markers with high correlation to the presence of mucosal healing constitute a cost-effective substitute to repeated endoscopies. Recent studies have reported that the prostaglandin E-major urinary metabolite (PGE-MUM) level was significantly higher in the active phase of patients with ulcerative disease (UC) than those in the remission phase. In the active UC phase, the stimulation of inflammatory cytokines, such as tumor necrosis factor-α, leads to the upregulation of cyclooxygenase-2 (COX-2) leading to PGE2 secretion in mucosal tissue. PGE2 plays an important role in the progression of inflammation. A precise measure of serum PGE2 is difficult due to the short half-life of PGE2 in the blood. Conversely, the urinary metabolite of prostaglandin E-major (PGE-MUM, 7-hydroxy-5,11-diketotetranor-prosta-1,16-dioic acid) is stable and may reflects the histological severity of inflammation. The aim of this concept study is to evaluate the PGE-MUM concentration in urine of patients with IBD in parallel with the standard investigation of Calprotectin in stool and to assess if urinary PGE-MUM should be able to serve as a simple and robust substitutive biomarker for the non-invasive evaluation of the inflammation of the mucous membrane tissues. The measurement of PGE-MUM in urine could give patients with IBD more comfort than the measurement of calprotectin in stool.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) include Crohn's disease (CD) and ulcerative colitis (UC) are chronic inflammations of the digestive tract with periods of remission of variable duration. As the timing of relapse is unpredictable, and current monitoring is symptoms-based, there remains a window between the initial upregulation of the inflammatory response and the onset of clinical symptoms at which point the inflammatory episode is well established. Endoscopy displays direct evidence of mucosal injury but as means of predicting relapse is not suitable for regular use. Biological examinations are looking for signs of inflammation such as the presence of inflammatory anemia or thrombocytosis, frequently found, or increased C-reactive protein (CRP), a nonspecific marker poorly correlated with endoscopic inflammation; or looking for signs of malabsorption such as hypoalbuminemia or vitamin deficiencies. These serum markers are limited in fulfilling the role as a prognostic marker of relapse.

The best non-invasive biomarker compared to endoscopic examination for the monitoring of IBD is the fecal calprotectin (CF). Calprotectin is a 36 kiloDalton, calcium- and zinc-binding protein that comprises up to 60% of cytosolic proteins in neutrophils, being released during apoptosis or necrosis. Its fecal concentration is therefore proportional to neutrophilic influx into the intestinal tract, which is a feature of active IBD. FC is therefore an accurate surrogate marker of active endoscopic disease in IBD patients, its sensitivity is between 70% - 100%, with a specificity of 44% - 100%, depending on the threshold value used. FC measurement is now widely available and is being incorporated into routine clinical practice. The advantages of fecal biomarkers are that samples (feces) are easy to obtain, can be collected at home, can be serially obtained, and can be relatively easy to analyze with the sample posted to the laboratory for analysis.

Point-of-care urinary markers can represent interesting candidates as tools for monitoring inflammatory activity in IBD and for assessing the risk of imminent disease flares. According to the latter concept, clinical remission should be paired with biological and endoscopic evidence of mucosal inflammatory inactivity in IBD patients. Expressed in ratio to creatinine, the more complicated collection of 24 hours urine is useless.

Recent studies have reported that prostaglandin E2 (PGE2) is produced in the mucosa of the intestine of areas affected by IBD and the PGE2 plays important role in the progression of inflammation. In the active UC phase, the stimulation of inflammatory cytokines, such as tumor necrosis factor-α, leads to the upregulation of cyclooxygenase-2 (COX-2) leading to PGE2 secretion in mucosal tissue. In blood, PGE2 is immediately metabolized by 15-hydroxy prostaglandin dehydrogenase (15-PGDH), which is present in the lung and colon, into 15-keto-PGE2. Next, in the liver and kidney, 15-keto-PGE2 is converted into 13,14-dihydro-15-keto PGE2 by the action of Δ13-reductase, followed by β-oxidation and ω-oxidation; this is finally converted to PGE-MUM (7α-hydroxy-5,11-diketotetranor-prosta-1,16-dioic acid) and excreted along with urine. A precise measure in the blood of PGE2 was considered difficult due to the short half-life of PGE2 in the blood. Conversely, the urinary metabolite of prostaglandin E-major (PGE-MUM, 7-acid 5-hydroxy, 11-diketotetranor-prosta-1, 16-dioecious) is stable.

A correlation was reported (Arai, 2014) between PGE-MUM and inflammatory activity in IBD using the 3 severity score indexes - clinical, colonoscopic, and histological - Simple clinical colitis activity index (SCCAI), Mayo endoscopic scoring and Matts grading respectively (. When the cutoff value was set to 17 mg/g creatinine to distinguish Matts 1 from Matts 2-5, the sensitivity (equals to specificity), positive predictive value, negative predictive value, and accuracy of PGE-MUM were 0.82, 0.67, 0.93, and 0.83, respectively, compared with 0.69, 0.49, 0.93, and 0.69 for CRP respectively. The odds ratio was of 35 for the differentiation between cases in remission and active cases.

There is currently no study comparing urinary PGE-MUM and FC, which is the most validated and consensus biomarker of inflammation of the intestinal mucosa in Western countries. The proposed study aims to evaluate the correlation and bias between these two methods. The target population will be adult patients followed for chronic inflammatory bowel disease (IBD) diagnosed with certainty as Crohn's disease (CD) or ulcerative colitis (UC). The subjects will be recruited by specialized doctors in gastroenterology, IBD and nutrition assistance, on a voluntary basis after information and consent. These are patients benefiting from the usual IBD management circuit, either in outpatient for regular follow-up or hospitalized in case of recurrence for care aiming to limit the symptoms and duration of the acute inflammatory, and for whom a prescription for the measurement of fecal calprotectin and blood markers are required in routine care.

This proof-of-concept study might be used to direct future clinical validation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 60 years
* Patients with chronic inflammatory bowel disease, IBD (Crohn's or Ulcerative colitis)
* Patients with active or inactive disease (remission)
* Patients treated as part of their routine care and required to undergo a routine blood test, fecal tests and endoscopic examination, if applicable
* Patients covered by the social security scheme and / or professional health insurance
* Patients giving their free and informed consent after information

Exclusion criteria :

* Patients who have been deemed unfit to participate in the study by the attending physician
* Patients under 18 years
* Patients who have undergone colorectal surgery with complete resection or who have undergone intestinal resection surgery within six months
* Patients taking irritating laxatives, nonsteroidal anti-inflammatory drugs (NSAIDs) and drug formulations containing prostaglandins at the time of urine collection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with inflammatory bowel disease (IBD or UC) consulting, for the follow-up of their chronic disease, the gastroenterology department of Beaujon Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Correlation between urinary PGE-MUM and fecal Calprotectin concentrations | 12 months
  A statistical analysis will allow to evaluate the correlation and bias between urinary PGE-MUM concentration in mg/g-creatinine and fecal calprotectin concentration in patients with chronic inflammatory bowel disease (IBD). To compare the urinary PGE-MUM level equivalence according to predetermined calprotectin values recognized as biological cut-points, e.g. Calprotectin <50μg /g-stool is considered normal; > 250μg /g-stool is considered active inflammation.

SECONDARY OUTCOMES:
Correlation between urinary PGE-MUM and serum CRP concentrations | 12 months
  A statistical analysis will allow to evaluate the correlation and bias between urinary PGE-MUM concentration and serum C-reactive protein (CRP;mg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de biochimie clinique - Hôpital Beaujon, Clichy, France